CLINICAL TRIAL: NCT04111029
Title: Assessment of Response to Locoregional Therapy Using Liquid Biopsy in Patients With Hepatocellular Carcinoma
Brief Title: Liquid Biopsy in Hepatocellular Carcinoma
Acronym: HCCGenePanel
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Madhumita Premkumar, Assistant Professor, Department of Hepatology, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: INT/HEP/1078
Record Dates: First submitted 2019-09-26; First posted 2019-10-01 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Hepatic Carcinoma Malignant Primary Non-Resectable
Keywords: Hepatocellular carcinoma; Cell Free tumor DNA; Liquid Biopsy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Noninvasive Prenatal Testing; Liquid Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cell free DNA in Plasma will be stored
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Unresectable HCC undergoing locoregional therapy: Patients with unresectable HCC who have no curative option like tumour ablation, resection or transplantation and are being taken for locoregional therapy will be recruited
  Interventions: Diagnostic Test: Cell Free DNA

INTERVENTIONS:
Diagnostic Test: Cell Free DNA — Pre and post procedure plasma cell free DNA will be assessed for response to locoregional therapy
  Other Names: Liquid biopsy

SUMMARY:
Circulating tumor DNA (ctDNA) carrying tumor-specific sequence alterations has been found in the cell-free fraction of blood. Hepatocellular carcinoma (HCC) specimens are difficult to obtain, and noninvasive methods are required to assess cancer progression and characterize underlying genomic features. Use of 'liquid biopsy' by assessing circulating cell free DNA enables the clinician to offer targeted immunotherapy or signaling pathway inhibitors. It also offers a model to prove response to locoregional or immunotherapy therapy and predict tumor recurrence non-invasively.

DETAILED DESCRIPTION:
Novelty:

Mutation analysis may not only help identify cancer drivers, but they can also provide useful data to predict response to other treatment modalities such as immunotherapies, particularly immune checkpoint blockade. There is published data on liquid biopsy in India from oncology in the field of pulmonary and renal cancers, but these studies have not been done in cirrhosis or in HCC patients.

Objectives In this project we hope to develop a biomarker panel which helps us prognosticate patients and tailor targeted therapy as per their genetic mutation landscape. The treatment options for advanced HCC are limited, and tissue biopsy is not routinely performed.

Methods In this pilot project, we will analyze 30 patients with unresectable hepatocellular carcinoma, ineligible for liver transplantation, who will undergo locoregional therapy in the form of transarterial chemoembolization (TACE) or radioembolization (TARE) for tissue diagnosis of tumor tissue DNA and circulating tumor DNA. We will design personalized assays targeting somatic rearrangements of each tumor to quantify serum ctDNA. Exome sequencing will be performed using cell-free DNA and paired primary tumor tissue DNA in order to create a non-invasive liquid biopsy for diagnosis and prognostication of HCC.

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular carcinoma BCLC stages B and C of all aetiology, unresectable
* Age 18-70 years of either sex

Exclusion Criteria:

* Contemplating Hepatic resection or OLT
* Refractory ascites
* Severe Coagulation disorders prior to the procedure (PTI <70% and Platelet count < 80,000/mm3)
* Hepato-Renal syndrome
* Chronic Kidney Disease
* Acute decompensation like Hepatic encephalopathy and variceal bleeding
* Any known malignancy other than HCC
* Life expectancy < 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A) All new consecutively diagnosed cases of Hepatocellular carcinoma (HCC) fulfilling the inclusion criteria, presenting to the Hepatology OPD and admitted to the LICU and/or wards for loco-regional therapy for the first time.
  * All new cases of HCC diagnosed as per the AASLD 2018 guideline. HCC will be staged according to the Barcelona Clinic Liver Cancer (BCLC- Staging) system.
  * The patients undergoing their first LRT (TACE/TARE/SBRT) with or without Sorafenib for HCC who are not eligible for resection/ liver transplantation or any other curative modality.
  * Treatment allocation, as per the updated BCLC staging system and treatment strategy, which is also endorsed by the AASLD guidelines for the management of HCC
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-01-16 (Actual); Primary Completion 2023-12-16 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Comparison of exome sequencing of primary tumor tissue and cell-free DNA from plasma samples | 0, 90 days
Serial Quantification of ctDNA in plasma samples by means of real-time PCR post treatment | 90 days

SECONDARY OUTCOMES:
Time to first recurrence (local or distant) diagnosed on follow up dynamic imaging. | 90 days
Mortality | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Radhika Srinivasan, MD PhD, Study Chair — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, Choose Any State/Province, India

IPD SHARING:
Plan to Share IPD: Undecided